CLINICAL TRIAL: NCT02893670
Title: Tailored Re-evaluation for Adolescents With Inflammatory Bowel Disease in Transition (TRANSIT) Trial
Brief Title: Tailored Transition for IBD Adolescents
Acronym: TRANSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRANSIT01
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — X-Rays; Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored re-evaluation (Other): Radiologic (MRE) or endoscopic (sigmoidoscopy) evaluation:
  Following enrollment each patient will undergo a structured re-evaluation and transition process which will include radiologic intervention (MRE) for Crohn's patients and endoscopic intervention (sigmoidoscopy) for UC patients
  Interventions: Procedure: Radiologic (MRE) or endoscopic (sigmoidoscopy) evaluation

INTERVENTIONS:
Procedure: Radiologic (MRE) or endoscopic (sigmoidoscopy) evaluation — All patients will be assessed for drug levels and metabolites. Patients diagnosed with ileal or ileo-colonic crohn's will undergo an MR Enterography (MRE). In crohn's patients, MRE was shown to have a higher impact on patient management than colonoscopy. Patients diagnosed with either UC, IBD-U or Crohn's colitis will undergo a flexible sigmoidoscopy.
  Following re-evaluation each patient will undergo 2 transition meetings with pediatric and adult gastroenterologist as well as a meeting with IBD nurses and social worker.

SUMMARY:
Background: Smooth transition of adolescent patients diagnosed with inflammatory bowel diseases (IBD) to adult care is necessary in order to secure continues clinical management and to prevent possible deleterious clinical and psychosocial implications. In recent years there is an emphasis on successful transition, however, there are no standardized models or consensus guidelines incorporating both clinical and psychosocial aspects of transition. Objectives: To examine the effect a comprehensive clinical and psychosocial transition package on clinical management and patients outcomes in adolescents with IBD. Design: A prospective, trans-sectional study. Setting: The Schneider Children's Medical Center and the Rabin Medical Center. Participants: Children 17 year to 18 years who are diagnosed with IBD and are planned to initiate transition process to adult care. Main outcome measures: Change in clinical management as a result of tailored re-evaluation as a part of tailored transition package. Secondary outcome measures: a. The effect of a tailored transition package on patients' self-efficacy perception and readiness for transition. b. The effect of a tailored transition package on patient's outcomes (disease activity, flares, hospitalizations) during the first year following transition.

DETAILED DESCRIPTION:
General intervention scheme:

Patients with an established diagnosis of IBD (crohn's disease, ulcerative colitis or IBD-unclassified) will be enrolled between the age of 17 and 17.5 years. Patients are eligible for enrollment 6 months following diagnosis and onward.

Following enrollment each patient will undergo a structured re-evaluation as follows:

Each patient will be thoroughly examined and have height ,weight, body mass index performed as well as comprehensive laboratory examinations. Fecal sample for fecal calprotectin will be obtained as well. Extent of disease will be registered using the Montreal classification. Disease activity indices will be calculated according to the Harvey-Bradshaw Index (HBI) for crohn's and Partial Mayo Score (PMS) for UC.

Serum of patients treated with biologic medications will be analyzed for drug trough levels and anti-drug antibodies. Patients treated with thiopurines will have their blood analyzed for thiopurines metabolites. Patients will complete a "self-efficacy" and Transition Readiness Assessment Questionnaire (TRAQ). Both questionnaires were linguistically validated by bi-directional translation. Patients diagnosed with ileal or ileo-colonic crohn's will undergo an MR Enterography (MRE). In crohn's patients, MRE was shown to have a higher impact on patient management than colonoscopy. Patients diagnosed with either UC, IBD-U or Crohn's colitis will undergo a flexible sigmoidoscopy. Flexible sigmoidoscopy was recently shown to have a high degree of correlation with complete colonoscopy in assessments of UC activity.

Treating physicians are entitled to offer the patient a more extensive endoscopic evaluation (complete colonoscopy, gastroscopy) or radiologic evaluation (pelvic MRI, liver ultra-sound) if deemed necessary according to clinical indications.

Following the completion of clinical, laboratory and endoscopic/imaging evaluation a re-evaluation visit with both treating pediatric gastroenterologist and receiving adult gastroenterologist will be set. During this visit physicians will discuss the current treatment plan with the patient and the need for changes in therapeutic regimens (including step-up, step-down, adding or withdrawing optional treatments).

A transition visit with both treating gastroenterologists will be set 3-6 months following the re-evaluation visit (around 18 years of age) in order to assess the efficacy of the therapeutic plan and to complete the transition process. During the transition visit patients will, again, complete a "self-efficacy" and TRAQ questionnaires. In between the reevaluation visit and the transition visit the patients will be followed according to clinical indications by the treating pediatric gastroenterologist.

Prior to the transition visit each patient and parents will perform a transition preparation meeting with a multi-disciplinary team including a pediatric IBD nurse, an adult IBD nurse and a social worker. During this meeting the team will discuss practical issues concerning transition, instruct the patient on subjects specifically related to disease implications during late adolescence and early adulthood (substance abuse, alcohol, contraceptives, pregnancy, high education, work) and address special psycho-social needs/concerns. According to the team discretion, if a need for a meeting with the institute's psychologist is necessary, such meeting will be set within 30 days.

At 12 months following transition data on disease activity and outcomes including flares, hospitalizations and surgical interventions since transition will be collected. Data will be compared with an "historic" cohort of matched patients (case-controlled) who completed routine transition in the time period prior to the study in which transition was performed following 1-2 visits of the patient with both pediatric and adult gastroenterologists.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of inflammatory bowel disease
2. Age: 17 - 18 years ( inclusive)
3. Informed consent

Exclusion Criteria:

1. Recent diagnosis (last 6 months)

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in therapeutic regimen as a result tailored clinical re-evaluation at the end of the transition process | 6 months following enrollment

SECONDARY OUTCOMES:
The change in "self-efficacy" score at the end of the transition process | 6 months following enrollment
Disease activity (evaluated by crohn's disease activity index for crohn's and Mayo Clinic Index of Activity for UC) at 12 months following transition | 12 months following transition
The rate of flares during the first year following transition | 12 months following transition
The rate of hospitalizations during the first year following transition | 12 months following transition
Surgical rate during the first year following transition | 12 months following transition

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, MD, Study Chair — Tel Aviv University
Locations (1):
- Schenider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No